CLINICAL TRIAL: NCT04265820
Title: Prospective Clinical Study of Unilateral or Bilateral Implantation of Intraocular Lens in Cataract Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20191126
Record Dates: First submitted 2019-11-26; First posted 2020-02-12 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Cataract
Keywords: unilateral cataract; binocular functional vision; Multifocal Intraocular Lenses
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): The unilateral cataract patients in the Group 1 will undergo phacoemulsification and unilateral implantation of IOLs.The subjects will be divided into three subgroups according to the type of the IOLs.
  Interventions: Device: unilateral implantation of IOL
- Group 2 (Active Comparator): The bilateral cataract patients in the Group 2 will undergo phacoemulsification and bilateral implantation of IOLs.The subjects will be divided into three subgroups according to the type of the IOLs.
  Interventions: Device: bilateral implantation of IOL

INTERVENTIONS:
Device: unilateral implantation of IOL — unilateral phacoemulsification and implantation of IOL.IOL may be monofocal,bifocal ,or trifocal，according to the patients preference and the eyes condition.
  Arms: Group 1
Device: bilateral implantation of IOL — bilateral phacoemulsification and implantation of IOL.IOL may be monofocal,bifocal ,or trifocal，according to the patients preference and the eyes condition.
  Arms: Group 2

SUMMARY:
This is to evaluate the satisfaction of patient and postoperative functional vision of unilateral or bilateral Implantation of intraocular lens（IOLs） in cataract patients.

DETAILED DESCRIPTION:
The subjects will undergo uneventful phacoemulsification and implantation of IOL.

The subjects will be divided into two groups . The unilateral cataract patients in the Group 1 will undergo unilateral surgery, and the bilateral cataract patients in the Group 2 will undergo bilateral surgery. IOL may be monofocal,bifocal ,or trifocal，according to the patients preference and the eyes condition. In each group, the subjects will be divided into three subgroups according to the type of the IOLs.Compare binocular functional vision and the satisfaction of patient between the two groups at postoperative 3 months.Compare binocular functional vision and the satisfaction of patient with different IOLs among the subgroups.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unilateral or bilateral age related cataracts
* Regular corneal topography and Preoperative corneal astigmatism ≤ 0.75 Diopter

Exclusion Criteria:

* Pregnant or nursing women
* In the presence of other ocular diseases that may affect the stability of the lens capsule (pseudoexfoliation syndrome, glaucoma, traumatic cataract, Marfan syndrome, etc.)
* Pupil abnormality (non-reactive pupil, tonic pupils, abnormally shaped pupils, etc.)
* History of any clinically significant retinal pathology or ocular diagnosis (e.g. diabetic retinopathy, ischemic diseases, macular degeneration, retinal detachment, optic neuropathy optic nerv atrophy, amblyopia, strabismus, microphthalmos, aniridia, epiretinal membrane etc.) in the study eyes that could alter or limit final postoperative visual prognosis.
* Patients with history of ocular trauma or prior ocular surgery including refractive procedures
* postoperative visual acuity of worse than 0.2 logMAR in any eye
* Patients using systemic or ocular medication that affect visual acuity.
* Patients participating in other clinical trials during the study.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-10-28 (Actual); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
monocular and binocular visual acuity | 3 months postoperatively
  uncorrected distance visual acuity (UCVA), intermediate visual acuity, near visual acuity will be measured at 5m, 80cm and 40cm respectively. All visual acuity measurements will be conducted under photopic conditions (85 cd/m2) and at 100% contrast

SECONDARY OUTCOMES:
Binocular Contrast sensitivity | 3 months postoperatively
  Contrast sensitivity measures will be conducted binocularly, under photopic, mesopic (5 cd/m2), photopic with glare and mesopic with glare conditions, with the OPTEC 6500 contrast sensitivity test (Stereo Optical, USA). Contrast sensitivity will be evaluated at five spatial frequencies (1.5, 3, 6, 12, and 18 cycles per degree [cpd]). Patients will be allowed 5 minutes to adapt to each illumination level before testing.
Binocular Defocus Curve | 3 months postoperatively
  Binocular defocus curves will be obtained in all patients, positioned at 5m under photopic (>85 cd/m 2 ) condition to measure the visual acuity with each defocus lens, representing the consecutive visual function of each eye. Negative lenses were added in 0.50 D steps and the visual acuity will be recorded for each type of defocus level. The procedure will be then repeated but with positive lenses. The range of defocus evaluated is from -4.00D to +2.00D.
stereopsis | 3 months postoperatively
  Use block diagram of random-spot synoptophore to observe long distance stereopsis vision and yan's stereogram to observe short distance stereopsis vision.
Fusion function | 3 months postoperatively
  The fusion function of perception and movement (convergence and divergence)will be examined with a synoptophore.
Subjective visual quality | 3 months postoperatively
  Photic phenomena (score according to severity,0~4, higher scores mean worse)and spectacle dependence percentages will be evaluated by questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Qi Hong, PhD，MD, Study Director — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No